CLINICAL TRIAL: NCT02817048
Title: Thoracoscopic Surgery Without Chest Tube Placement in Patients With Peripheral Lung Nodules: A Prospective Randomized Trial
Brief Title: Tubeless VATS for Peripheral Lung Nodule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201603030RIND
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Solitary Pulmonary Nodule
MeSH Terms: conditions — Solitary Pulmonary Nodule | interventions — Chest Tubes; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tubeless (Active Comparator): Interventions: VATS without chest tube placement
  Interventions: Procedure: VATS without chest tube placement
- Chest tube (Active Comparator): VATS with chest tube placement
  Interventions: Device: chest tube; Procedure: VATS with chest tube placement

INTERVENTIONS:
Device: chest tube
  Arms: Chest tube
Procedure: VATS without chest tube placement — Patient received Video-Assisted Thoracic Surgery (VATS) wedge resection for peripheral lung nodule without chest tube placement (Tubeless)
  Arms: Tubeless
Procedure: VATS with chest tube placement
  Arms: Chest tube

SUMMARY:
Chest tube placement after thoracoscopy surgery had been generally accepted as routine procedure for removal of the residual intrapleural fluid and air, however, it would cause post-operative pain, prohibit ambulation after surgery, and prolong the hospital stay. According to the recent studies, omission of chest tube placement after minor thoracoscopic procedures (such as pulmonary wedge resection) had been safe and feasible, and it also reduced the post-operative pain and shortened the hospital stay. We will conduct a prospective randomized trial in National Taiwan University Hospital.

DETAILED DESCRIPTION:
We will enroll 100 patients with peripheral lung nodule who will be randomly assigned to no chest tube placement (tubeless group) or chest tube placement (control group) after thoracoscopic wedge resection with out without lymph adenectomy. The primary endpoints are to compare the post-operative hospital stay and post-operative pain sale between the two groups. The secondary endpoints are to compare the intercostal neuralgia and wound satisfaction one month after surgery between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* CT revealed peripheral lung nodule, with both size and depth less than 2 cm
* Aged 20 to 80 years

Exclusion Criteria:

* Patients with ventilatory defect
* Previous ipsilateral thoracic surgery
* Bleeding tendency or anticoagulant use
* Comorbidity including congestive heart failure, liver cirrhosis, chronic renal disease
* Pregnancy or breast feeding
* Immunocompromised or long-term steroid use
* Severe infected patient
* Patient who can not sign permit

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | 1 week

SECONDARY OUTCOMES:
Postoperative pain score | 1 week
Postoperative intercostal neuralgia | 1 month
Postoperative wound satisfaction | 1 month

OTHER OUTCOMES:
Hospital cost | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Study Director — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pompeo E, Mineo D, Rogliani P, Sabato AF, Mineo TC. Feasibility and results of awake thoracoscopic resection of solitary pulmonary nodules. Ann Thorac Surg. 2004 Nov;78(5):1761-8. doi: 10.1016/j.athoracsur.2004.05.083. PMID 15511470
- [Result] Rocco G, Romano V, Accardo R, Tempesta A, La Manna C, La Rocca A, Martucci N, D' Aiuto M, Polimeno E. Awake single-access (uniportal) video-assisted thoracoscopic surgery for peripheral pulmonary nodules in a complete ambulatory setting. Ann Thorac Surg. 2010 May;89(5):1625-7. doi: 10.1016/j.athoracsur.2010.01.087. PMID 20417792